CLINICAL TRIAL: NCT02461758
Title: Randomized Trial of High Dose vs. Standard Dose Influenza Vaccine in Inflammatory Bowel Disease Patients
Brief Title: Trial of High Dose vs. Standard Dose Influenza Vaccine in Inflammatory Bowel Disease Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2015-0813; Influenza in IBD (Other: Study Team)
Record Dates: First submitted 2015-05-26; First posted 2015-06-03 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Inflammatory Bowel Disease (IBD)
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Control Group (Other): A group of 20 healthy individuals without IBD, other chronic diseases, or immunosuppressive therapy will be enrolled. All healthy individuals will receive standard dose influenza vaccine SDIV.
  Interventions: Biological: Standard dose Influenza vaccine (SDIV)
- Vedolizumab Group + standard dose influenza vaccine (SDIV) (Other): A group of 20 patients who are currently on vedolizumab. All individuals in this group will receive SDIV
  Interventions: Biological: Standard dose Influenza vaccine (SDIV)
- High dose influenza vaccine (HDIV) (Other): This arm will be a double blind randomized controlled trial of High dose influenza vaccine (HDIV) for IBD patients on TNF monotherapy.
  40 patients will be enrolled and randomized in a 5:3 fashion to HDIV or SDIV. Randomization will generated by a random number generator and investigator will be blinded to randomization scheme.
  Interventions: Biological: High dose influenza vaccine (HDIV)
- Standard dose influenza vaccine (SDIV) (Other): This arm will be a double blind randomized controlled trial of standard dose influenza vaccine (SDIV) for IBD patients on TNF monotherapy.
  40 patients will be enrolled and randomized in a 5:3 fashion to HDIV or SDIV. Randomization will generated by a random number generator and investigator will be blinded to randomization scheme.
  Interventions: Biological: Standard dose Influenza vaccine (SDIV)

INTERVENTIONS:
Biological: Standard dose Influenza vaccine (SDIV)
  Arms: Control Group; Standard dose influenza vaccine (SDIV); Vedolizumab Group + standard dose influenza vaccine (SDIV)
Biological: High dose influenza vaccine (HDIV)
  Arms: High dose influenza vaccine (HDIV)

SUMMARY:
Inflammatory bowel disease (IBD) is a chronic inflammatory disorder of the gastrointestinal tract which includes Crohn's disease (CD) and ulcerative colitis (UC). A recent epidemiological investigation estimates that nearly 4 million people worldwide are affected and approximately 1.4 million of these cases occur in the United States. IBD can lead to debilitating symptoms, hospitalizations, decreased quality of life, frequent procedures and/or surgery. Treatment options consist of immunosuppressive therapy, such as systemic corticosteroids, immunomodulators (thiopurines and methotrexate) and/or biologics, such as tumor necrosis factor alpha (TNF) agents or an integrin inhibitor, vedolizumab. They can achieve clinical remission and decrease the risk of complications, but also increase the risk for opportunistic infections, including influenza.

Multiple studies have shown lower influenza vaccine responses in patients with IBD compared to healthy individuals; IBD patients treated with TNF agents or combination therapy (TNF inhibitors and immunomodulators) are very likely to mount a poor immune response. Influenza serum antibody concentration correlates with protection from infection following vaccination. Therefore, increasing influenza antibody responses in patients with IBD would appear to be critical to improving protection from influenza. A high dose (HD) influenza vaccine containing four times more hemagglutinin was licensed based on its ability to induce higher antibody concentrations compared to standard dose (SD) in adults 65 years or older.

ELIGIBILITY:
CASES Specific Aim #1 Inclusion Criteria

* A history of chronic (greater than 3 month) ulcerative colitis or Crohn's disease diagnosed and documented by the standard clinical, radiographic, endoscopic and histopathologic criteria.
* Ages 18-64
* Currently taking anti-TNF therapy (infliximab, golilumab, adalimumab, or certolizumab) for at least 3 months
* Exclusion Criteria
* Received season's influenza vaccine
* Allergy to eggs or influenza vaccine
* Currently use of systemic steroids in the past 3 months

Specific Aim #2 Inclusion criteria

* A history of chronic (greater than 3 month) ulcerative colitis or Crohn's disease diagnosed and documented by the standard clinical, radiographic, endoscopic and histopathologic criteria.
* Ages 18-64
* Currently on vedolizumab therapy

Exclusion Criteria

* Received season's influenza vaccine
* Allergy to eggs or influenza vaccine
* Currently use of systemic steroids in the past 3 months

Control group Inclusion criteria

* Age 18-64
* Willing to participate in study

Control group Exclusion criteria

* Currently on immunosuppressive therapy
* Has a chronic health condition that may have an impact on vaccine antibody concentrations as deemed by the investigators, including chronic liver disease, celiac disease, history of solid organ or bone marrow transplantation.
* Older than age 65 years
* Unconfirmed Measles, Mumps, and Rubella (MMR) vaccination status
* Patients in whom venipuncture are not feasible due to poor tolerability or lack of easy access.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2016-10; Primary Completion 2018-06 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Freddy Caldera, Principal Investigator — University of Wisconsin School of Medicine and Public Health, Madison
Locations (1):
- University of Wisconsin Hospital & Clinics, Madison, Wisconsin, United States

REFERENCES:
- [Result] Caldera F, Hillman L, Saha S, Wald A, Grimes I, Zhang Y, Sharpe AR, Reichelderfer M, Hayney MS. Immunogenicity of High Dose Influenza Vaccine for Patients with Inflammatory Bowel Disease on Anti-TNF Monotherapy: A Randomized Clinical Trial. Inflamm Bowel Dis. 2020 Mar 4;26(4):593-602. doi: 10.1093/ibd/izz164. PMID 31504526

RESULTS

PARTICIPANT FLOW:
Groups:
- Vedolizumab Group: A group of 20 patients who are currently on vedolizumab. All individuals in this group will receive SDIV
Period: Overall Study
Arm/Group | Control Group | Vedolizumab Group | High Dose Influenza Vaccine (HDIV) | Standard Dose Influenza Vaccine (SDIV)
Started | 20 | 20 | 26 | 15
Completed | 20 | 19 | 25 | 15
Not Completed | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Vedolizumab Group | High Dose Influenza Vaccine (HDIV) | Standard Dose Influenza Vaccine (SDIV) | Total
Number analyzed (Participants) | 20 | 19 | 25 | 15 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.35 (9.89) | 36.57 (16.16) | 34.96 (12.92) | 39.35 (11.98) | 37.81 (12.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 9 | 5 | 36
  Male | 10 | 7 | 16 | 10 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 19 | 19 | 25 | 14 | 77
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 19 | 25 | 15 | 79

OUTCOME MEASURES:

1. Primary Outcome: Measure Antibody Concentrations in Immunosuppressed IBD Patients Who Receive High Dose and Standard of Care Dose Influenza Vaccine
Description: Influenza vaccine antibody concentration will be measured in immunosuppressed IBD patients who receive high dose and standard of care dose influenza vaccine.
  Higher antibody concentrations are associated with better protection from infection.
Time Frame: Pre-immunization and 2-4 weeks post immunization
Measure: Median (Inter-Quartile Range); unit: Antibody Titer
Groups:
- High Dose of Influenza Vaccine (HDIV) Group: This arm will be a double blind randomized controlled trial of high dose influenza vaccine (HDIV) for IBD patients on TNF monotherapy.
  40 patients will be enrolled and randomized in a 5:3 fashion to HDIV or SDIV. Randomization will generated by a random number generator and investigator will be blinded to randomization scheme.
- Standard Dose Influenza Vaccine (SDIV) Group: This arm will be a double blind randomized controlled trial of standard dose influenza vaccine (SDIV) for IBD patients on TNF monotherapy.
  40 patients will be enrolled and randomized in a 5:3 fashion to HDIV or SDIV. Randomization will generated by a random number generator and investigator will be blinded to randomization scheme.
Arm/Group | High Dose of Influenza Vaccine (HDIV) Group | Standard Dose Influenza Vaccine (SDIV) Group | Vedolizumab Group | Control Group
Number analyzed (Participants) | 25 | 15 | 19 | 20
Antibody Titer
  Influenza A H1N1, pre-immunization | 160 [80 to 240] | 160 [80 to 160] | 160 [80 to 320] | 160 [80 to 160]
  Influenza A H1N1, 2-4 weeks post immunization | 320 [150 to 320] | 160 [80 to 320] | 320 [160 to 640] | 320 [160 to 320]
  Influenza A H3N2, Pre-immunization | 80 [40 to 160] | 40 [20 to 40] | 80 [80 to 160] | 80 [40 to 80]
  Influenza A H3N2, 2-4 weeks post immunization | 160 [80 to 320] | 80 [40 to 160] | 320 [160 to 320] | 160 [160 to 160]
  Influenza B Victoria,Pre-immunization | 10 [10 to 20] | 10 [10 to 20] | 20 [10 to 20] | 20 [20 to 35]
  Influenza B Victoria, 2-4 weeks post immunization | 20 [15 to 20] | 20 [20 to 40] | 20 [20 to 40] | 20 [20 to 40]
  Influenza B Yamagata, Pre-immunization | 10 [10 to 20] | 10 [10 to 20] | 20 [10 to 40] | 20 [10 to 35]
  Influenza B Yamagata, 2-4 weeks post immunization | 10 [10 to 20] | 20 [10 to 20] | 40 [20 to 40] | 20 [13 to 40]

2. Secondary Outcome: Response Rate Against Influenza Vaccine in Patients With Inflammatory Bowel Disease: Number of Participants Positive for Seroconversion
Description: Vaccine response rates for influenza vaccines in patients with inflammatory bowel disease will be accessed by number of patients who has shown significant seroconversion. Seroconversion is defined as a four fold increase in antibody concentration from preimmunization to 4 weeks post immunization.
Time Frame: 4 weeks
Measure: Number; unit: participants
Groups:
- High Dose of Influenza Vaccine(HDIV) Group: This arm will be a double blind randomized controlled trial of high dose influenza vaccine (HDIV) for IBD patients on TNF monotherapy.
  40 patients will be enrolled and randomized in a 5:3 fashion to HDIV or SDIV. Randomization will generated by a random number generator and investigator will be blinded to randomization scheme.
- Contorl Group: A group of 20 healthy individuals without IBD, other chronic diseases, or immunosuppressive therapy will be enrolled. All healthy individuals will receive standard dose influenza vaccine SDIV.
Arm/Group | Standard Dose Influenza Vaccine (SDIV) Group | High Dose of Influenza Vaccine(HDIV) Group | Vedolizumab Group | Contorl Group
Number analyzed (Participants) | 15 | 25 | 19 | 20
participants
  Influenza A H1N1 | 1 | 9 | 4 | 4
  Influenza A H3N2 | 6 | 11 | 7 | 6
  Influenza B Victoria | 1 | 4 | 2 | 0
  Influenza B Yamagata | 0 | 0 | 1 | 0
  At least one virus | 7 | 15 | 9 | 7
  At least two viruses | 1 | 7 | 3 | 3
  Three viruses | 0 | 2 | 1 | 0

3. Secondary Outcome: Seroprotection: Number of Participants With Antibody Concentration at Least 1:40 at Week 4 Postimmunization
Description: Seroprotection is defined as an antibody concentration of at least 1:40 at 4 weeks post-immunization which confers protection from infection in about 50% of individuals
Time Frame: 4 weeks
Measure: Number; unit: participants
Groups:
- Standard Dose Influenza Vaccine (SDIV) Group: This arm will be a double blind randomized controlled trial of standard dose influenza vaccine (SDIV) for IBD patients on TNF monotherapy.
  40 patients will be enrolled and randomized in a 5:3 fashion to HDIV or SDIV. Randomization will generated by a random number generator and investigator will be blinded to randomization scheme.
  .
Arm/Group | Standard Dose Influenza Vaccine (SDIV) Group | High Dose of Influenza Vaccine(HDIV) Group | Vedolizumab Group | Control Group
Number analyzed (Participants) | 15 | 25 | 19 | 20
participants
  Influenza A H1N1 | 15 | 25 | 19 | 20
  Influenza A H3N2 | 15 | 25 | 19 | 20
  Influenza B Victoria | 8 | 6 | 10 | 10
  Influenza B Yamagata | 6 | 6 | 11 | 8
  At least one virus | 15 | 25 | 19 | 20
  At least two virus | 15 | 25 | 19 | 20
  Three viruses | 8 | 9 | 13 | 11

4. Secondary Outcome: Seroprotection: Number of Participants With Antibody Titer of 160 at Week 4 Post-immunization
Description: Seroprotection is defined by the FDA as post-immunization concentration of 1:160 that confers protection from infection to 95% of the population.
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Standard Dose Influenza Vaccine (SDIV) Group | High Dose of Influenza Vaccine(HDIV) Group | Vedolizumab Group | Control Group
Number analyzed (Participants) | 15 | 25 | 19 | 20
participants
  Influenza A H1N1 | 12 | 24 | 19 | 18
  Influenza A H3N2 | 6 | 21 | 16 | 17
  Influenza B Victoria | 0 | 0 | 0 | 0
  Influenza B Yamagata | 0 | 0 | 1 | 0
  At least one virus | 13 | 25 | 19 | 20
  At least two virus | 5 | 20 | 16 | 15
  Three viruses | 0 | 0 | 1 | 0

5. Secondary Outcome: Measure Antibody Concentrations in Immunosuppressed IBD Patients Who Receive High Dose and Standard of Care Dose Influenza Vaccine
Description: as for outcome 1
Time Frame: 6 months post-immunization
Measure: Median (Inter-Quartile Range); unit: Antibody Titer
Arm/Group | High Dose of Influenza Vaccine (HDIV) Group | Standard Dose Influenza Vaccine (SDIV) Group | Vedolizumab Group | Control Group
Number analyzed (Participants) | 25 | 15 | 19 | 20
Antibody Titer
  Influenza A H1N1, 6 months post immunization | 160 [80 to 320] | 160 [80 to 320] | 160 [160 to 320] | 160 [80 to 320]
  Influenza A H3N2, 6 months post immunization | 80 [40 to 80] | 80 [40 to 160] | 160 [80 to 160] | 80 [80 to 160]
  Influenza B Victoria, 6 months post immunization | 20 [10 to 20] | 20 [18 to 40] | 40 [20 to 40] | 20 [20 to 40]
  Influenza B Yamagata, 6 months post immunization | 20 [10 to 20] | 20 [10 to 20] | 20 [20 to 40] | 20 [20 to 40]

ADVERSE EVENTS:
Time Frame: Up to 7 days
Description: AEs were recorded after administration of the vaccine from days 0-6 using the adverse event dairy. Adverse event data is reported for 24 participants in the HDIV arm as 1 participant did not submit the diary card for adverse event reporting. Adverse event are reported just for anti-TNF monotherapy group HDIV and SDIV since these were the primary outcome.No AEs were collected for vedolizumab group and control group as they were secondary outcomes which were dependent on primary outcomes.
Arm/Group | High Dose Influenza Vaccine (HDIV) | Standard Dose Influenza Vaccine (SDIV)
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/15
Other Adverse Events (participants affected / at risk) | 13/24 | 8/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Influenza Vaccine (HDIV) (N=24) | Standard Dose Influenza Vaccine (SDIV) (N=15)
Local reactions: Pain (Skin and subcutaneous tissue disorders) | 10 (10) | 4 (4)
Local reaction: Redness (Skin and subcutaneous tissue disorders) | 7 (7) | 5 (5)
Swelling (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5)
fever (General disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 9 (9) | 5 (5)
Muscle Aches (General disorders) | 12 (12) | 8 (8)
Arthralgia (General disorders) | 6 (6) | 4 (4)
Fatigue (General disorders) | 13 (13) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-01-27): https://cdn.clinicaltrials.gov/large-docs/58/NCT02461758/Prot_000.pdf
  • Statistical Analysis Plan (2015-08-13): https://cdn.clinicaltrials.gov/large-docs/58/NCT02461758/SAP_001.pdf